CLINICAL TRIAL: NCT05273996
Title: Phenotype Predictors of Cognitive Outcomes in Geriatric Depression
Brief Title: Predictors of Cognitive Outcomes in Geriatric Depression
Acronym: NBOLD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: David Steffens (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, David Steffens, Samuel "Sy" Birnbaum/Ida, Louis and Richard Blum Chair in Psychiatry Professor and Chair, Department of Psychiatry, UConn Health
Organization: UConn Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IE-13-048H-6.1; R01MH108578 (NIH)
Record Dates: First submitted 2021-12-13; First posted 2022-03-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder; Neuroticism; Cognitive Change; Stress
Keywords: Late Life Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline; Bupropion; Desvenlafaxine Succinate

STUDY DESIGN:
Intervention Model Description: Naturalistic study using FDA approved antidepressants to examine the effects of stress and neuroticism on outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Depressed (Other): Subjects receive FDA-approved antidepressants
  Interventions: Drug: Sertraline, bupropion, desvenlafaxine

INTERVENTIONS:
Drug: Sertraline, bupropion, desvenlafaxine — Study geriatric psychiatrists prescribe FDA-approved antidepressants using a treatment algorithm consistent with the STAGED (Duke Somatic Treatment Algorithm for Geriatric Depression) approach, with standardization of treatment in the first six months beginning with sertraline, with the option of augmentation with bupropion or switch to desvenlafaxine. Beyond six months of acute treatment, subjects are treated based on the study psychiatrist's clinical assessment and recommendations, consistent with STAGED guidelines.
  Other Names: Zoloft; Wellbutrin; Pristiq

SUMMARY:
This study will focus on examining effects of stress on long-term mood and cognitive outcomes of late-life depression. It will also example the neural underpinnings of these changes using structural and functional brain imaging. Understanding how effects of stress in older depressed adults, as well as factors that might minimize those effects, lead to particular mood and cognitive outcomes will inform future development of novel prevention strategies.

DETAILED DESCRIPTION:
In this renewal of R01MH108578, the investigators are seeking to extend findings from the initial study to focus on effects of stress in longitudinal mood and cognitive outcomes of late-life depression (LLD) and to examine stress effects on brain structure and function in LLD. Severe or persistent stressors can result in a number of behavioral and mood changes, including anxiety, dysphoric mood, sleep disruption, altered appetite, and withdrawal from social and pleasurable activities. These stress-related consequences are particularly salient when considering longitudinal outcomes of treated LLD. They may be compounded by an individual's longstanding maladaptive patterns of response to stress, embodied in the construct of neuroticism, which the investigators have shown to be related to poor mood and cognitive LLD outcomes. Moreover, Andreescu et al. (2019) introduced a model of depression recurrence that incorporates the homeostatic disequilibrium hypothesis, which proposes that in geriatric remitted depression, neural networks are in fragile homeostasis that is threatened by stress exposure. Networks of particular importance in stress of LLD outcome are the Default Mode Network (DMN), Salience Network (SN) and Executive Control Network (ECN).

The Neurobiology of Late Life Depression (NBOLD) study began enrolling older depressed and never depressed controls in 2013, enrolling 132 depressed and 44 controls, and currently follows 77 depressed and 22 controls. Subjects are well characterized in terms of mood, cognition, personality and stress (including specific measures obtained during the present COVID pandemic). It is well suited to examine stress effects on longitudinal mood and cognitive outcomes. For the renewal, the study will follow current subjects and recruit 75 new subjects, who will be followed for up to 5 years with annual cognitive testing, stress measures and baseline and two-year functional brain magnetic resonance imaging (fMRI) scan.

In this renewal, the investigators will examine the following specific aims:

1. To study effects of stressors (obtained on a variety of measures) and neuroticism on longitudinal mood and cognitive outcomes in older adults with history of major depressive disorder (MDD).
2. To study effects of stress and neuroticism on brain structure and function in older adults with MDD history.
3. To explore relationships among variables in Aims 1 and 2 with longitudinal multivariable statistical models.

ELIGIBILITY:
Inclusion Criteria:

* major depression, single episode or recurrent;
* ability to read and write English;
* Mini-Mental State Examination >25.

Exclusion Criteria:

* lifetime alcohol/drug dependence
* conditions associated with brain abnormalities such hydrocephalus, benign and cancerous brain tumors, epilepsy, Parkinson's disease, Huntington's chorea, dementia, demyelinating diseases, etc.
* untreated endocrine disorder other than diabetes mellitus
* established clinical diagnosis of dementia
* other primary psychiatric disorders, e.g., panic disorder, social phobia, obsessive- compulsive disorder, schizoaffective disorder, schizophrenia, bipolar disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRAS) | Three years
  Measure of depression severity and Recurrence of Depression Minimum Score = 0; Maximum Score = 60; Higher score means worse outcome
Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Neuropsychological Battery Total Score | Three years
  Global cognitive measure; Minimum Score = 0; Maximum Score = 100; Higher score means better outcome
Cognitive clinical diagnosis | three years
  Participant records will be reviewed annually by the consensus panel. The study will convene a panel of experts to review each case, including the PI, treating geriatric psychiatrists and study neuropsychologist. Panel members review the following information for each participant: 1) initial evaluation and most recent clinical depression study notes, 2) neuropsychological testing profiles, 3) informant report of cognitive decline based on the Dementia Severity Rating Scale, 4) study structural MRI images to determine vascular burden, and 5) additional neurological and clinical neuropsychological consultations when available. The panel discusses the case until a consensus cognitive diagnosis is reached.

SECONDARY OUTCOMES:
Functional brain magnetic resonance imaging (fMRI) scan changes in resting state functional connectivity. | Two years
  A change in the strength of connectivity within a network and between two networks will be determined by comparing the strength of connectivity at baseline and at two years. The functional connectivity strength is reflected by a z score of normalized Pearson correlation coefficient using the Fisher transformation.
Functional brain magnetic resonance imaging (fMRI) scan structural imaging changes | Two years
  Measures from structural imaging in the key brain regions will be the volumetric measurement from T1-weighted MRI. A change in the volume of a brain structure will be determined by subtracting the regional volume at baseline from two years.

OTHER OUTCOMES:
Neuroticism subtest score on NEO Personality Inventory | Three years
  Neuroticism domain and its subdomains will be examined; Minimum Score = 0; Maximum Score = 92; Higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: David Steffens, M.D., M.H.S., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This R01 will develop important new data on 75 subjects. These data will be available to investigators both within UConn and outside the institution.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: Potential investigators will gain knowledge of the project through NIH Reporter and through Dr. Steffens' UConn webpage. They will be able to contact Dr. Steffens and he will work with the investigator to determine the nature of what the investigator wishes to study to ensure that he/she has a complete data set that will allow for a successful analysis. Dr. Steffens' team will create an anonymized data set, encrypt it, and electronically transfer it to the investigator.
  Dr. Steffens will maintain a list of approved analyses and track progress of manuscripts and publications. In addition, consistent with National Institute of Mental Health (NIMH)requirements, Dr. Steffens will plan to submit data via the NIMH Data Archive (NDA).